CLINICAL TRIAL: NCT07261735
Title: Three-Dimensional Evaluation of Wear and Clinical Survival of Attachments Reproduced With Customized Composites for Clear Aligner Therapy: A Prospective Observational Clinical Study
Brief Title: Clinical Evaluation of Customized Attachment Composites in Clear Aligner Therapy
Status: Recruiting | Type: Observational
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Sponsor
Other Study IDs: SBU-GULHANE-ORTHO-ATTACH-2025
Record Dates: First submitted 2025-11-21; First posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-08

CONDITIONS: Clear Aligner Therapy - Attachment Wear and Bonding Performance
Keywords: Clear aligner therapy; Orthodontic attachments; Split-mouth design; Customized composites; Surface wear; Clinical survival

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group 1: All Participants: All participants receive four different composite materials using a randomized split-mouth design. Each quadrant is assigned one composite for attachment reproduction
  Interventions: Device: GC G-ænial A'Chord Universal Composite; Device: Spectra ST HV (High Viscosity); Device: Spectra ST LV (Low Viscosity); Device: GC Aligner Connect Composite

INTERVENTIONS:
Device: GC G-ænial A'Chord Universal Composite — Universal composite resin used as the control material for attachment reproduction.
Device: Spectra ST HV (High Viscosity) — High-viscosity universal composite resin clinically used for clear aligner attachment reproduction.
Device: Spectra ST LV (Low Viscosity) — Low-viscosity universal composite resin clinically used for clear aligner attachment reproduction.
Device: GC Aligner Connect Composite — Customized composite resin specifically developed for clear aligner attachments.

SUMMARY:
This prospective observational clinical study aims to evaluate the three-dimensional surface wear and clinical survival of orthodontic attachments fabricated with customized composite materials used in clear aligner therapy. Attachments play a critical role in the biomechanical efficiency of aligner treatment by facilitating planned tooth movements. However, the mechanical and surface properties of the composites used for attachment fabrication may affect their wear behavior and long-term stability.

In this study, four different composite materials will be tested using a split-mouth design in patients treated with clear aligners. Each quadrant will receive a different composite, including both customized and universal types. All attachments will be fabricated using standardized digital templates and bonded under identical clinical conditions. Surface wear will be evaluated using three-dimensional optical scanning and metrology software at baseline, 1 week, 1 month, 3 months, and 6 months. Lost attachments will be replaced and recorded but excluded from wear analysis.

The results of this study are expected to provide valuable insights into the optimal material selection for clear aligner attachments, improving treatment accuracy and clinical durability.

DETAILED DESCRIPTION:
The study is a prospective, observational, split-mouth clinical investigation conducted at the University of Health Sciences, Gülhane Faculty of Dentistry, Department of Orthodontics. It aims to compare the surface wear resistance and clinical performance of attachments fabricated with different composite resins used in clear aligner therapy.

Four composite materials will be evaluated: GC G-ænial A'Chord (control), Spectra ST HV, Spectra ST LV, and GC Aligner Connect. Each patient will receive four different materials applied to separate quadrants following a randomized split-mouth allocation. The study planning and randomization were performed by a single researcher to ensure methodological consistency. All attachments will be fabricated using standardized digital templates based on the virtual treatment plan. The bonding procedure will be carried out by one investigator using Transbond XT adhesive and 37% phosphoric acid etching for 15 seconds.

Intraoral scanning will be performed at baseline, 1 week, 1 month, 3 months, and 6 months. The scanned data will be analyzed using Zeiss Inspect software to quantify volumetric and surface wear. All 3D alignments and superimpositions will be performed by a blinded evaluator to ensure objectivity. Lost or fractured attachments will be recorded and replaced but excluded from quantitative wear analysis.

All participants will be followed for six months. Statistical analysis will include repeated-measures ANOVA and post-hoc testing with a significance level of p < 0.05. Reliability will be evaluated using the intraclass correlation coefficient (ICC).

This study has been approved by the Gülhane Scientific Research Ethics Committee of the University of Health Sciences (Approval No: 2024/015, August 19, 2025). The findings are expected to enhance understanding of how different composite materials influence attachment wear and longevity in clear aligner therapy, thereby improving the accuracy and clinical predictability of treatment outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Fully erupted permanent dentition.
* No existing prosthetic restorations.
* Mild-to-moderate dental crowding or spacing (2-6 mm).
* Patients who are scheduled to undergo clear aligner therapy at the Department of Orthodontics, Gülhane Faculty of Dentistry, between 01.08.2025 and 01.08.2026.
* Patients who agree to participate and provide informed consent.

Exclusion Criteria:

* History of previous fixed orthodontic treatment.
* Patients with poor predicted compliance or low cooperation.
* Presence of severe or generalized periodontal disease.
* High caries incidence or untreated caries.
* Poor oral hygiene
* Habitual consumption of hard foods.
* Bruxism
* Congenitally missing permanent teeth.
* Dental developmental anomalies.
* Teeth with existing composite resin restorations or ceramic crowns on buccal surfaces (which may interfere with attachment bonding or wear analysis)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study population consists of individuals with fully erupted permanent dentition who are beginning clear aligner treatment at the Gülhane Faculty of Dentistry. Participants are enrolled prospectively after providing written informed consent for participation and for additional follow-up intraoral scans used for attachment wear analysis. Eligible patients present with mild-to-moderate crowding or spacing, show adequate oral hygiene and periodontal health, and have no prosthetic restorations or history of fixed orthodontic treatment. Patients with bruxism, high caries activity, generalized periodontal disease, poor cooperation, or buccal-surface restorations are excluded. As part of routine orthodontic care, all participants receive standardized oral hygiene instructions, including a daily tooth-brushing protocol and recommendations for toothbrush and toothpaste selection. No invasive or non-routine procedures are performed.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2025-08-25 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
3D Surface Wear of Orthodontic Attachments | Baseline to 6 months
  The three-dimensional surface wear of attachments will be evaluated using Zeiss Inspect software (Zeiss GmbH) by comparing baseline (T0) and follow-up scans (T1: 1 week, T2: 1 month, T3: 3 months, T4: 6 months). Wear will be quantified as total surface deviation (sigma) across the entire attachment surface and as point deviations measured at predefined corner and mid-surface points. All 3D alignments and analyses will be performed by an independent, blinded examiner who is unaware of the composite allocation for each quadrant.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Health Sciences, Gülhane Faculty of Dental Medicine, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to the inclusion of identifiable intraoral scans, photographs, radiographs, and clinical records that cannot be fully de-identified. In addition, national data protection regulations prohibit the external sharing of personal health information. Only aggregated study results will be made available through scientific publications.